CLINICAL TRIAL: NCT01279304
Title: Radiotherapy After Primary CHEMotherapy for cT1-2cN1M0 Breast Cancer.: a Multicentre Prospective Registration Study.
Brief Title: Radiotherapy After Primary Chemotherapy for Breastcancer
Acronym: RAPCHEM
Status: Completed | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: The Netherlands Cancer Institute (Other); Diakonessenhuis, Utrecht (Other)
Responsible Party: Sponsor
Other Study IDs: 10-04-10/02
Record Dates: First submitted 2011-01-17; First posted 2011-01-19 (Estimated); Last update posted 2022-10-14 (Actual); Status verified 2014-02

CONDITIONS: Breast Cancer
Keywords: breast cancer; locoregional recurrence rate; neoadjuvant chemotherapy and surgery; radiotherapy; risk model; overall survival; relapse free survival; cT1-2cN0-1 breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1. Low risk: 1. Surgical strategy is full axillary lymph node dissection after primary systemic treatment and in case of:
     a. all nodes negative: ycN0
     or
  2. Surgical strategy is sentinel node procedure only performed prior to primary systemic treatment and in case of:
     a. only micrometastases in the SN, and no risk factors (grade 3, LVI, tumour size > 3 cm)
     or
  3. Surgical strategy is sentinel node procedure only performed after primary systemic treatment and in case of:
     1. no metastases in the post chemo SN
  Interventions: Radiation: radiation - no radiation see intervention description
- Group 2: Intermediate risk: 1. Surgical strategy is full axillary lymph node dissection after primary systemic treatment and in case of:
     a. 1-3 nodes positive: ypN1
     or
  2. Surgical strategy is sentinel node procedure only performed prior to primary systemic treatment and in case of:
     1. micrometastases in the SN and at least 1 risk factor; or
     2. ≤ 2 macrometastases and no risk factor
     or
  3. Surgical strategy is sentinel node procedure only performed after primary systemic treatment and in case of:
     1. micrometastases in the post chemo SN and no risk factors (grade 3, LVI, tumour size > 3 cm)
  Interventions: Radiation: radiation: see intervention description
- Group 3. High risk: 1. Surgical strategy is full axillary lymph node dissection after primary systemic treatment and in case of:
     a. 4 or more nodes positive: ypN2
     or
  2. Surgical strategy is sentinel node procedure only performed prior to primary systemic treatment and in case of:
     1. ≤ 2 macrometastases in the sentinel node prior to primary systemic treatment in the presence of risk factors like Grade 3, lymphangioinvasion, tumour size > 3 cm; or
     2. 3 macrometastases, 2 macrometastases and 1 micrometastase, 1 macrometastase and 2 micrometastases.
     or
  3. Surgical strategy is sentinel node procedure only performed after primary systemic treatment and in case of:
     1. Micrometastases in the post chemo SN, and at least one risk factor
     2. ≤ 3 macrometastases in the post chemo SN; or
     3. 2 macrometastases and 1 micrometastase, 1 macrometastase and 2 micrometastases
  Interventions: Radiation: radiation: see intervention description

INTERVENTIONS:
Radiation: radiation - no radiation see intervention description — after MRM in group 1 (low risk): no radiotherapy after BCT in group 1 (low risk): radiation treatment of the breast with boost (optional)
  Groups: Group 1. Low risk
Radiation: radiation: see intervention description — after BCT in group 2 (intermediate risk): radiation treatment of the breast with boost (optional) after MRM in group 2 (intermediate risk): radiation treatment of the thoracic wall If no full ALND is performed in group 2 (intermediate risk) add radiation treatment of level 1 and 2 of the axilla.
  Groups: Group 2: Intermediate risk
Radiation: radiation: see intervention description — after MRM in group 3 (high risk): radiation treatment of the thoracic wall and supraclavicular nodes after BCT in group 3 (high risk): radiation treatment of the breast with boost (optional) and supraclavicular nodes If no full ALND is performed group 3 (high risk) add radiation treatment of level 1 and 2 of the axilla.
  Groups: Group 3. High risk

SUMMARY:
The primary aim of the study is to evaluate the 5 yr locoregional recurrence rate (LRR) in cT1-2cN0-1(cytology/histology and/or positive SN, excluding patients with > 3 pathologic axillary nodes on imaging) breast cancer patients, treated with neoadjuvant chemotherapy, breast surgery, and radiotherapy that is protocolized based on the pathology findings after chemotherapy and definitive surgery (ypTNM stage).

DETAILED DESCRIPTION:
Primary systemic treatment for breast cancer patients used to be given only to patients with locally advanced disease. Although until now no studies have been reported that primary systemic treatment leads to a superior survival compared to adjuvant chemotherapy [Mauri et al, 2005; Mieog et al, 2007], the last years have been showing an increase in the use of primary systemic treatment , also for patients with earlier stages of breast cancer. The suggested advantages of this policy are 1) that primary systemic treatment allows for monitoring of the response on the treatment, such that the type of chemotherapy can be changed in case of no response, and 2) that primary systemic treatment may shrink the tumour volume, allowing for a higher percentage of breast conserving therapy [Mieog et al, 2007]; and 3) the overall 40% chance of converting positive axillary nodes pre-PST to negative, questioning the need for an axillary dissection [Fontein et al, 2013; Kuehn et al, 2013]. A major disadvantage of primary systemic treatment is however, that the indications for post-operative radiotherapy are based upon studies where loco-regional recurrences were correlated to the pathological T and N stage in patients who had not been treated with chemotherapy before surgery. Since primary systemic treatment is affecting the pathological T and N stage, the indications for post-operative radiotherapy in these patients have become uncertain.

Objective: The primary aim of the study is to evaluate the 5 yr locoregional recurrence rate (LRR) in cT1-2cN0-1(cytology/histology and/or positive SN, excluding patients with > 3 pathologic axillary nodes on imaging) breast cancer patients, treated with neoadjuvant chemotherapy, breast surgery, and radiotherapy that is protocolized based on the pathology findings after chemotherapy and definitive surgery (ypTNM stage). The secondary aim is to develop a risk model based on risk factors, that can be used to predict which of the patients with a cT1-2cN0-1 breast carcinoma, treated with neoadjuvant chemotherapy and surgery, have a 5 yr LRR > 8 % if radiotherapy is withheld.

Study design: This study is a multicentre prospective cohort study. Study population: In total 710 patients with cT1-2pN0-1, excluding ≥cN2 and patients with > 3 pathologic axillary nodes on imaging, breast cancer, treated with at least three cycles of chemotherapy followed by breast and axillary surgery are eligible for the study.

During 5 years (2011-2015) patients diagnosed for primary breast cancer and eligible according to the criteria will be registered by the National Cancer Registry in this project.

Currently, three surgical strategies are being followed in cT1-2N0-1 patients, treated with primary systemic treatment :

1. A full axillary lymph node dissection is performed after the primary systemic treatment , OR
2. A sentinel node procedure is carried out prior to neoadjuvant treatment, and no further axillary surgery is performed after chemotherapy, if the patient is clinically node negative (ycN0)), OR
3. A sentinel node procedure is carried out only after primary systemic treatment , in case patient is still/has become clinically node negative (ycN0).

For all three above mentioned strategies, patients are divided into three risk groups, mainly based on the post chemotherapy pathological nodal status (strategy 1 and 3), and on the pre-chemotherapy pathological nodal status and ycN0 status (strategy 2). In addition, for all three strategies the cT and the ycT status are taken into account to choose the recommended guideline.

The radiation treatment guidelines for the subsequent three risk groups consist of:

1. Group I - low risk (N = 237):

   1. after MRM: no radiotherapy
   2. after BCT: radiation treatment of the breast with boost (optional)
2. Group II - intermediate risk (N = 237):

   1. after MRM: radiation treatment of the thoracic wall
   2. after BCT: radiation treatment of the breast with boost (optional)
   3. if no full ALND is performed: add radiation treatment to level 1 and 2
3. Group III - high risk group(N = 237):

   1. after MRM: radiation treatment of the thoracic wall and supraclavicular nodes
   2. after BCT: radiation treatment of the breast with boost (optional), and supraclavicular nodes
   3. if no full ALND is performed (not recommended): add radiation treatment to the axilla level 1 and 2 RT of the axillary (after ALND) and internal mammary chain nodes is optional for group III, based on the local protocol. In case of a positive sentinel node in the internal mammary chain prior to chemotherapy, internal mammary chain irradiation is strongly recommended Main study parameters/endpoints: The primary endpoint is the 5 yr locoregional recurrence rate (LRR). Secondary endpoints are 10 year LRR, 5, 10, and 15 yr relapse free survival rates (all events except lost to follow-up, invasive contralateral cancer, and secondary primary (non-breast) invasive cancer) and overall survival rates. In addition, analyses will be performed to investigate whether pre-radiotherapy factors (e.g. like age < 40 yr, response to chemotherapy, tumour size) can be identified that correlate with a high LRR.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Currently no clear data are present in literature showing the indications for radiotherapy in this patient group. Based on literature that is available for patients treated with chemotherapy after surgery we have chosen what we think might be the optimal treatment from a benefit/risk perspective. The study focuses on adequate registration of all risk factors, treatment, and outcome.

Date amendment: 1 July 2013

The main reason for writing an amendment is that current guidelines on axillary treatment are changing, both with respect to surgery and with respect to radiation treatment. Not sufficient data are yet present in literature to define a sound evidence based guideline. However, recent new data strongly suggest that the guidelines should be adapted. Therefore, we adapted the guidelines within the framework of this protocol, with as aim to carefully follow and record the outcome of patients treated with these new guidelines. Whilst writing this amendment, we also used this opportunity to better define "suspicious nodes" on imaging, and to add another very relevant endpoint: relapse free survival.

ELIGIBILITY:
Inclusion criteria:

* cT1-2 invasive breast cancer, without or with one or more pathologically proven tumour positive axillary lymph nodes (either by sentinel node biopsy, ultrasound/palpation guided biopsy or fine needle aspiration)
* At least 3 cycles of primary systemic treatment have been given (irrespective of the regimen)
* No standard axillary lymph node dissection is performed prior to chemotherapy

Exclusion criteria:

* cT3-T4 invasive breast cancer prior to any treatment
* Patients with > 3 suspicious axillary nodes on imaging
* cN2-3 prior to any treatment
* More than focally irradical surgery and breast conserving therapy

To investigate whether a patient is eligible for the RAPCHEM study, a meticulous examination of the axilla is necessary. Therefore each patient should undergo an ultrasound of the axilla and if possible an ultrasound guided needle biopsy UNB (FNA or core). The US/UNB can be performed instantly or as second look in case of enlarged nodes on MRI. The criteria for performing an UNB are:

* Cortex >2.3 mm not measured at the poles of the node; or
* Disappearance of the fatty hilum; or
* Asymmetric bulging of the cortex of a lymph node;

If a PET-CT is performed the worst outcome of the two studies is accepted as the real clinical stage of the axilla (i.e. 1 PA proven positive lymph node on ultrasound and 3 on PET-CT; means 3 positive lymph nodes)

The N status of the axilla prior to chemotherapy is based upon:

* Positive PET-CT of more than one but less than 4 axillary nodes; since the specificity of PET positive nodes in a proven breast cancer patient is very high, pathology confirmation is not absolutely required
* Positive US of axillary nodes; at least one should be pathology proven tumour positive
* The worst outcome of 1 and 2 represents the most reliable clinical axillary staging.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with cT1-2cN0-1(cytology/histology and/or positive SN, excluding patients with > 3 pathologic axillary nodes on imaging) breast cancer, treated with at least three cycles of chemotherapy followed by breast surgery are eligible for the study.
Sampling Method: Probability Sample
Enrollment: 851 (Actual)
Dates: Start 2011-01; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
locoregional recurrence rate | 5 Yr
  to evaluate the 5 year locoregional recurrence rate (LRR) in cT1-2cN0-1(cytology/histology and/or positive SN, excluding patients with > 3 pathologic axillary nodes on imaging) breast cancer patients, treated with neo-adjuvant chemotherapy, breast surgery, and radiotherapy that is protocolised based on the pathology findings after chemotherapy and definitive surgery (ypTNM stage).

SECONDARY OUTCOMES:
risk model based on rick factors | 5 Yr
  to develop a risk model based on risk factors, that can be used to predict which of the patients with a cT1-2cN1 breast carcinoma, treated with neoadjuvant chemotherapy and surgery, have a 5 yr LRR > 8 % if radiotherapy is withheld.
10 year LRR | 10 Yr
  10 year Locoregional Recurrence Rate
5 Yr relapse free survival rate | 5 Yr
  5 year relapse free survival rate (all events except lost to follow-up, invasive contralateral cancer, and secondary primary (non-breast) invasive cancer).
10 yr relapse free survival rate | 10 Yr
  10 year relapse free survival rate (all events except lost to follow-up, invasive contralateral cancer, and secondary primary (non-breast) invasive cancer).
15 Yr relapse free survival rate (all events except lost to follow-up, invasive contralateral cancer, and secondary primary (non-breast) invasive cancer). | 15 Yr
  and 15 year relapse free survival rate (all events except lost to follow-up, invasive contralateral cancer, and secondary primary (non-breast) invasive cancer).
5 Yr overall survival rate | 5 Yr
  5 year overall survival rate
10 Yr overall survival rate | 10 yr
  10 year overall survival rate
15 Yr overall survival rate | 15 Yr
  15 year overall survival rate

CONTACTS AND LOCATIONS:
Overall Officials: L.J Boersma, Principal Investigator — Maastricht University Medical Centre; A Voogd, Principal Investigator — Maastricht University; R Houben, Principal Investigator — Maastricht University Medical Centre
Locations (6):
- Netherlands (6):
  - UMC St Radboud Nijmegen, Nijmegen, Gelderland
  - Maastro clinic, Maastricht, Limburg
  - Dr. B. Verbeeten Institute, Tilburg, North Brabant
  - The Netherlands Cancer Institute, Amsterdam, North Holland
  - Diakonessen Hospital Utrecht, Utrecht
  - UMC Utrecht, Utrecht

REFERENCES:
- [Background] Boersma LJ, Verloop J, Voogd AC, Elkhuizen PHM, Houben R, van Leeuwen AE, Linn S, de Munck L, Pijnappel R, Strobbe L, van Dalen T, Wesseling J, Poortmans P. Radiotherapy after primary CHEMotherapy (RAPCHEM): Practice variation in a Dutch registration study (BOOG 2010-03). Radiother Oncol. 2020 Apr;145:201-208. doi: 10.1016/j.radonc.2020.01.018. Epub 2020 Feb 10. PMID 32058873
- [Derived] de Wild SR, de Munck L, Simons JM, Verloop J, van Dalen T, Elkhuizen PHM, Houben RMA, van Leeuwen AE, Linn SC, Pijnappel RM, Poortmans PMP, Strobbe LJA, Wesseling J, Voogd AC, Boersma LJ. De-escalation of radiotherapy after primary chemotherapy in cT1-2N1 breast cancer (RAPCHEM; BOOG 2010-03): 5-year follow-up results of a Dutch, prospective, registry study. Lancet Oncol. 2022 Sep;23(9):1201-1210. doi: 10.1016/S1470-2045(22)00482-X. Epub 2022 Aug 8. PMID 35952707